CLINICAL TRIAL: NCT05158504
Title: The Effects of Motivational Messages Sent to Emergency Nurses During the COVID-19 Pandemic on Job Satisfaction, Compassion Fatigue, and Communication Skills: A Randomized Controlled Trial
Brief Title: The Effect of Motivational Messages on Emergency Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Hilal KARTAL, PhD student, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SBU-HAMIDIYE-KARTAL-00001-2021
Record Dates: First submitted 2021-11-15; First posted 2021-12-15 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Satisfaction; Compassion Fatigue; Communication, Social
MeSH Terms: conditions — Personal Satisfaction; Compassion Fatigue; Communication | interventions — Information Motivation Behavioral Skills Model

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivation (Experimental): Motivational notifications were sent to the nurses in the motivational group (n=30) via SMS messages to their mobile phones at 07.00, 12.00 and 16.00 for 21 days. Like a good morning message that allows you to start the day with a beautiful energy (Example: Thank you for the hard and selfless work you do every day. We love and appreciate angels like you and you. Good morning). Motivational notifications sent to the participants were prepared each day to be different from the previous day. Data were obtained with the Individual Introduction Form, Job Satisfaction, Compassion Fatigue and Communication Skills Scale.
  Interventions: Other: Motivation
- Control (No Intervention): Motivational notifications were not sent to the nurses in the control group (n=30) and they continued their routine work in the emergency room. only pretest and posttest were applied. Data were obtained with the Individual Introduction Form, Job Satisfaction, Compassion Fatigue and Communication Skills Scale.

INTERVENTIONS:
Other: Motivation — Motivational notifications were sent via SMS message to the nurses in the motivation group (n=30) at 07.00, 12.00 and 16.00 for 21 days.
  Arms: Motivation

SUMMARY:
Aim and objectives: The aim of this study is to examine the effect of motivational notifications applied to emergency nurses on job satisfaction, compassion fatigue and communication skills during the COVID-19 pandemic.

Background: Emergency room nurses working on the front lines during the COVID-19 pandemic; many factors such as excessive workload, prolonged working hours, threat of infection, death of the patients they care for have caused them to experience physical, social and psychological problems.

Design: It is a randomized controlled, open-label study. Methods: This study was carried out with a total of 60 nurses working in the emergency units of two training and research hospitals in Istanbul. Participants were divided into motivational group and control group. Motivational notifications were sent via Short Message Service (SMS) to the mobile phones of the participants in the motivational group (n=30) for 21 days. No motivational notification was sent to the control group (n=30) during this process. Data were obtained with the Individual Introduction Form, Job Satisfaction, Compassion Fatigue and Communication Skills Scale.

ELIGIBILITY:
Inclusion Criteria:The nurses working in the emergency room, working only in the day shift on weekdays, using mobile phones and volunteering to participate in the study were included in the study.

-

Exclusion Criteria: Exclusion criteria for the study included being on leave for any reason (maternity, annual, medical) during the study dates, not completely filling in the data collection forms, or withdrawing from the study.

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hilal KARTAL, Istanbul, Beylikdüzü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Motivation
Started | 32 | 33
Completed | 30 | 30
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivation | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.86 (7.56) | 28.70 (6.95) | 28.78 (7.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 14 | 17 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Education Level;High school,Associate degree,Undergraduate,Postgraduate [Count of Participants; unit: Participants]
  High school | 6 | 4 | 10
  Associate degree | 5 | 4 | 9
  Undergraduate | 10 | 18 | 28
  Postgraduate | 9 | 4 | 13
Professional Experience [Count of Participants; unit: Participants]
  <1 year | 2 | 7 | 9
  1-5 years | 8 | 7 | 15
  6-10 | 9 | 10 | 19
  ≥10 | 11 | 6 | 17
Time Working in Current Unit [Count of Participants; unit: Participants]
  <1 year | 3 | 8 | 11
  1-5 years | 12 | 13 | 25
  5-10 years | 11 | 7 | 18
  ≥10 | 4 | 2 | 6
Weekly Working Hours [Count of Participants; unit: Participants]
  <40 hours | 5 | 2 | 7
  >40 hours | 25 | 28 | 53
Feels the profession suits them [Count of Participants; unit: Participants]
  yes | 22 | 20 | 42
  none | 8 | 10 | 18
Intends to continue working [Count of Participants; unit: Participants]
  YES | 10 | 16 | 26
  NONE | 20 | 14 | 34

OUTCOME MEASURES:

1. Primary Outcome: Job Satisfaction-Short Scale
Description: Job satisfaction scale is in a 5-point Likert type and is graded as (1- Absolutely disagree and 5-Absolutely agree). Scoring of the scale is calculated as a minimum of 1 and a maximum of 5 points, and the average of 5 related items is taken. The lowest score that can be obtained from the scale is 5 and the highest score is 25. Accordingly, the decrease in the average score of the participants indicates that job satisfaction decreases; an increase in the average score indicates an increase in job satisfaction.
Time Frame: Baseline and after 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivation | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 17.70 (3.26) | 14.10 (3.77)

2. Primary Outcome: Compassion Fatigue-Short Scale
Description: The scale aims to measure secondary trauma and occupational burnout. Items are rated on a 10-point Likert-type scale ranging from rarely/never (1) to very often (10). The total possible score ranges from 13 to 130, with higher scores representing a higher level of compassion fatigue.
Time Frame: Baseline and after 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Motivation
Number analyzed (Participants) | 30 | 30
score on a scale | 54.53 (21.78) | 36.73 (12.43)

3. Primary Outcome: Communication Skills Scale
Description: This scale was developed to determine how people evaluate their own communication skills. It consists of 25 items on a 5-point Likert-type scale ranging from always (1) to never (5). The scale yields a score ranging from 25 to 125. High scores reflect a positive perception of the person's communication skills.
Time Frame: Baseline and after 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control: Motivational notifications were not sent to the nurses in the control group.
- Motivation: Motivational notifications were sent to the nurses in the control group.
Arm/Group | Control | Motivation
Number analyzed (Participants) | 30 | 30
score on a scale | 88.36 (15.37) | 100.93 (9.31)

ADVERSE EVENTS:
Time Frame: Three weeks.
Arm/Group | Control | Motivation
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Our results are limited to the participants in this study, and cannot be generalized to all nurses working in emergency units during the COVID-19 pandemic. The study spanned a relatively brief period, and messages have a short-term effect. Therefore, long-term studies with larger sample groups are needed to determine the long-term effectiveness of motivational messages. The participants could not be blinded due to the study design, and demoralization could limit the validity of the results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT05158504/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT05158504/SAP_001.pdf